CLINICAL TRIAL: NCT00495729
Title: A Single-blind, Randomised, Placebo-controlled, 15 Day Repeated-dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of SB-649868 and Its Interaction With the CYP3A4 Isoenzyme in Healthy Male Subjects.
Brief Title: 15-Day Repeated-Dose Study With SB-649868 And Its Interaction With CYP3A4 Isoenzyme In Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: OXS104092
Record Dates: First submitted 2007-06-29; First posted 2007-07-03 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: SB-649868,; Simvastatin; Repeated dose,
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Subjects in Cohort 1 will be randomized to receive 5 milligram (mg) of SB-649868 or Placebo along with 10 mg of simvastatin.
  Interventions: Drug: SB-649868; Drug: Placebo; Drug: Simvastatin
- Cohort 2 (Experimental): Subjects in Cohort 2 will be randomized to receive two or three times higher than the starting dose of SB-649868 or Placebo along with 10 mg of simvastatin.
  Interventions: Drug: SB-649868; Drug: Placebo; Drug: Simvastatin
- Cohort 3 (Experimental): Subjects in Cohort 3 will be randomized to dose higher than that administered in Cohort 2 of SB-649868 or Placebo along with 10 mg of simvastatin.
  Interventions: Drug: SB-649868; Drug: Placebo; Drug: Simvastatin

INTERVENTIONS:
Drug: SB-649868 — Subjects will receive SB-649868 5 mg, 25 mg tablets orally 1 hour prior to simvastatin administration.
Drug: Placebo — Subjects will receive matching placebo tablets to SB-649868 orally 1 hour prior to simvastatin administration.
Drug: Simvastatin — Subjects will receive Simvastatin 10 mg tablets orally.

SUMMARY:
Subjects will be screened within 28 days, Simvastatin dose and single SB-649868 dose 10 and 7 days prior to repeat dosing respectively, 15 days SB-649868 repeat dosing with safety and cognition function tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male subjects aged between 18 and 65 years of age inclusive.
* Body weight =50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive.
* Healthy as judged by responsible physician. No clinically significant abnormality identified on the medical or laboratory evaluation and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator and the Medical Monitor considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Subjects will have blood pressure measurements within the normal range for healthy volunteers.

Exclusion Criteria:

* The subject has a positive pre-study urine drug/ alcohol urine screen.
* A positive pre-study Hepatitis B surface antigen, Hepatitis C antibody, or HIV 1/2 result at the screening visit.
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units.
* Subject complains of sleep disturbances and/ or is receiving treatment for sleep disorders.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-04-18 (Actual); Primary Completion 2007-08-04 (Actual); Study Completion 2007-08-04 (Actual)

PRIMARY OUTCOMES:
-AE, Lab values and cardiovascular monitoring after the SD and 14 days RD period (15 days) | after the SD and 14 days RD period (15 days)
- SB649868 levels on days -7, 1, 4, 7 and 14 (pre-dose and post-dose) | on days -7, 1, 4, 7 and 14 (pre-dose and post-dose)
- Simvastatine and Beta-idroxy-simvastatine levels on days -10,1,4,7 and 15 | on days -10,1,4,7 and 15

SECONDARY OUTCOMES:
Cognitive functions, sleep profile and appetite assessment on days -7, 7 and 14. | on days -7, 7 and 14.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

REFERENCES:
- See also: Results for study OXS104092 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/OXS104092?search=study&search_terms=OXS104092#rs